# Phase IIb Study of the Efficacy of FLU-v, a Broad Spectrum Influenza Vaccine in an H1N1 Influenza Healthy Human Challenge Model

# **Informed Consent Form**

NCT Number: NCT03180801

**EudraCT Number:** 2016-002134-74

Last date of approval: January 2018

Version: Final v3.2\_31JAN2017



# INFORMED CONSENT FORM

Phase IIb Study of the Efficacy of Flu-v, a Broad Spectrum

Protocol Title Influenza Vaccine in an H1N1 Influenza Healthy Human

Challenge Model

**Sponsor:** PepTcell Limited (t/a SEEK)

Protocol number: FLU-v-004

**Protocol version:** Final v2.2\_31JAN2017

**EudraCT Number:** 2016-002134-74

SEEK

Central Point,

Sponsor's address: 45 Beech Street,

London,

EC27 8AD

Research Ethics

Committee (REC) Ref:

16/NE/0227

Principal

Investigator: Dr Andrea Guerra

**Research sites:** hVIVO Services Limited sites at:

Queen Mary BioEnterprises Innovation Centre

(1) 42 New Road, London E1 2AX, UK

Telephone: 0207 756 1414 Manchester Science Parks

(2) Kilburn House, Lloyd Street North, Manchester M15 6SE, UK

Telephone: 0161 402 3470

Dr Jeremy Dennison

Pharmacy and Clinical services

(3) Hammersmith Medicines Research Ltd

Cumberland Avenue, London, NW10 7EW, UK

Telephone: 0208 961 4130

# 1 Invitation and instructions for filling in this form

We are inviting you to take part in a research investigation (a clinical study). Please read this information sheet before you decide whether to take part. If you have any questions, please ask a member of staff.

# 2 Why we are doing this research

The purpose of this research is to test the effects of an experimental drug in the form of a vaccine called FLU-v (the "study vaccine"). PepTcell (the 'Sponsor') is developing this vaccine to prevent people getting infected with Influenza. The vaccine is 'experimental' because regulatory authorities (such as the Medicines and Healthcare products Regulatory Agency in the UK) have not approved it for use in patients

To test new vaccines, we first give the vaccine and then subsequently try to infect healthy volunteers 6 weeks later with a virus in a quarantined residential facility to see if the vaccine can help in preventing the infection. In this research, the virus we will use is a live strain of Influenza (the 'study virus'), which has been prepared to the highest standards by the National Institutes of Health in the US. hVIVO has given various Influenza viruses to over 1000 research participants in the past and the study virus has been given to over 185 volunteers in the past.

Up to 123 participants will be receiving the study virus in this research study. The Sponsor is paying hVIVO Services Limited ('hVIVO') to carry out this research. hVIVO will be paid by the sponsor to




# **INFORMED CONSENT FORM**

perform the study on their behalf.

We will use various procedures to collect blood, nasal swabs and other samples in order to measure the effects of the study vaccine and the study virus on the body, particularly your nose and blood cells, before, during and after viral infection.

Samples and information may be used for current and future ethically approved research. Samples may also be used to develop and test our laboratory methods and the equipment that we use.

#### 2.1 About Influenza

Influenza is an infectious disease commonly referred to as 'the flu'. The Influenza virus is easily spread by coughs and sneezes, and can cause mild to severe illness. Influenza illness is often confused with the common cold, but is caused by a different virus and the symptoms are usually worse than a cold. People who have influenza may have fever, chills, cough, sore throat, runny or stuffy nose, muscle or body aches, headaches, and tiredness. Some may also have vomiting and diarrhoea, although this is more common in children. Certain people, (e.g., the elderly, pregnant women, very young children and people with certain chronic health conditions [e.g., asthma, heart failure]) are particularly vulnerable to influenza and can become very ill and some may develop life-threatening complications such as severe lung infections, sinus and ear infections.

Influenza viruses tend to change from year to year, and may cause seasonal outbreaks in a single country (an epidemic) or worldwide (a pandemic); pandemics can result in millions of deaths. The approved treatments for flu are drugs called zanamivir and oseltamivir, but new drugs are needed because the flu virus may be becoming 'resistant' to these drugs. If the flu virus becomes resistant to a drug, the drug will not be as effective against flu as it may have been in the past.

Vaccines can protect people from infection with Influenza, but they are targeted to specific types ('strains') of Influenza virus, which may or may not be circulating in the population during a particular seasonal flu epidemic.

#### 2.2 About Flu-v

Flu-v (the 'study drug') is being developed for the prevention and reduction in symptoms of multiple types (Broad-spectrum) of Influenza virus infection. Given as a vaccine (an injection in to your upper arm), it works by stimulating the cells of immune system to fight the virus. It also contains water and an additional substance known as ISA-51, which is an adjuvant, which helps the body produce a stronger defence response. The study vaccine will be given as either 1 or 2 injections in to your upper arm. FLU-v plus adjuvant will now be referred to as the 'study vaccine' from hereon in.

In order to further test the effectiveness and safety of the study vaccine at 1 or 2 doses, healthy volunteers will be exposed to the study virus once they have received their allocated treatment.

# 3 Are there any health benefits?

The study vaccine is aiming to protect against a broad range of flu types. Since study vaccine is still under research, taking part will not improve your health, although you may develop some resistance to some of the various types of Influenza.

# 4 What am I being asked to do?

This information describes what is involved in the 'clinical trial' you have been asked to consent to.




# **INFORMED CONSENT FORM**

hVIVO conducts these clinical trials in small groups of participants using a variety of research procedures (described in **Section 8**) to study if the experimental vaccine works. You will be asked to consent to the research procedures on the 'Consent form' at the end of this document.

As our research progresses, the types and timings of research procedures that will be used in the study may differ, but standard procedures will be used to closely monitor your safety and wellbeing whilst you are participating.

# 5 Do I have to take part?

No, taking part is entirely voluntary. We invited you because you said you wanted to be in a clinical trial, but you can still decide not to take part. If you do take part, you can leave at any time without saying why and without penalty or loss of any of the benefits to which you were entitled (see **Section 13**). However, if we have already given you the study virus, we will advise you to stay in the Quarantine Unit until you are no longer considered infectious. If we have already given you the study vaccine we will advise you to come for 1 or 2 follow-up safety visits to ensure you remain well.

If you decide or need to leave the study for whatever reason we would ask you to inform and discuss your decision, if possible, with your study staff as soon as possible.

# 6 What should I do if I want to take part?

Please read all the information carefully before you decide whether or not to take part. You should ask the staff any questions you have, and then when you are ready, sign the form at the end of this information sheet. You will then have some tests, including blood and urine tests, to see if you are suitable for this study. We will give you a copy of your signed and dated consent form and the clinical trial visit schedule.

To be suitable for the study, you must be healthy, aged 18 to 55 years, have a low resistance to Influenza (measured by a blood test), and meet the study rules for entry. The study staff must think you are suitable and your General Practitioner (GP) or doctor will also be contacted and asked to provide details of your medical history from at least the last 2 years. There may be some costs associated with obtaining your medical history from your GP which hVIVO will pay for in full.

We will look after you during the study and check your health as necessary. If the staff wants to double check a test result, he/she may ask you to return for this extra test.

# 7 The Study Process

Up to 123 participants (or 'volunteers') will be enrolled to receive the study virus after they have been given the 2 injections of the study vaccine (treatment groups discussed in section 7.2). To achieve this we will enrol up to 168 participants to ensure we invite the required number to the quarantine facility. Each participant will be in the study for about 5 months from screening to their last clinic visit and in the hVIVO medical unit (i.e. Quarantine) for approximately 10 days. Please see the study design diagram below.

The procedures and tests required for this study are shown in the study Visit Schedule at the end of this information sheet.


Version: Final v3.2 31JAN2017



# INFORMED CONSENT FORM Study Design Diagram



# 7.1 Visit 1: Screening

It is important that you are in good health. We will take blood and urine samples and do a number of procedures and tests to check that you are suitable. These are described in **Section 8**.

We will ask you about your medical history and any medicines and treatments you have been taking. You must answer honestly and fully.

You may not be able to take part if any of your blood or urine results are abnormal (outside of the normal range), and you may be asked to provide an additional sample for repeat testing. If an abnormal result is medically significant, we will advise you to consult your GP.

In addition to safety blood assessments, your blood will be tested for Hepatitis types A, B and C viruses (which affect your liver), and Human Immunodeficiency Virus (HIV- the virus that causes Acquired Immune Deficiency Syndrome [AIDS]). If any of these tests are positive, you will not be able to take part in the study.

People can be infected with hepatitis viruses and/or HIV and not know about it. If you are infected with these viruses, this can affect the types of jobs you can do, and any health insurance or life assurance policies that you have. If you think you could be infected, or you do not want to be tested, speak to the study staff. We will keep your test results and anything you tell us confidential. If you are infected, you will be invited to attend for counselling and a further consultation, and if you wish, the study doctor will inform your GP and arrange for you to see a specialist.

If you have ever had a Herpes infection (e.g., cold sores or genital Herpes), there is a small possibility that this infection could return after you have been given the study virus. We have seen this on very rare occasions in previous studies, and it should resolve quickly. You must inform the study doctor if you currently have an active Herpes infection, or have had one in the last 30 days.




# **INFORMED CONSENT FORM**

# 7.2 Visit 2 and 3: Administration of the vaccine

If you are invited to attend the vaccination visit, you may be asked to attend the hVIVO unit to give a screening (pre-vaccination) blood sample prior to the first planned vaccination visit (Day -43). You may be reimbursed for reasonable time and travel expenses for this visit, at hVIVOs discretion.

You will be admitted to the Hammersmith Medicines Research Unit in London on Day -43 and Day - 22. When you arrive at the Hammersmith Unit, we will check to ensure you remain healthy and eligible to continue on the study to receive the study vaccine.

You will be allocated at random (by chance – like tossing a coin) to one of 3 study treatment groups:

- 1 2 doses of placebo injection
- 2 the study vaccine and a placebo injection 21 days later, or
- 3 the study vaccine (FLU-v) and the same again in 21 days.

You will therefore have a 2 in 3 chance of receiving either 1 or 2 doses of the study vaccine. A placebo is a dummy drug that looks exactly like the study drug, but contains none of the active ingredients. The staff looking after you over the course of the study will not be aware of the treatment group you have allocated to unless we need to for safety purposes. By comparing the 3 treatment groups it can then be seen if one treatment group is more effective and / or safer than another.

At each visit we will provide you with diary cards that you will have to fill in at home for 3 weeks after each injection. These diary cards will help us understand if you are unwell after receiving a study vaccine.

# 7.3 Visit 4: Quarantine stay

Once you have received your 2 allocated study vaccines and you remain well, we will invite you to our Quarantine unit in London on Day -2 or Day -1, 1 or 2 days before you are given the study virus on Day 0. When you arrive at the Quarantine Unit on Day -2 or Day -1, we will check to see if you are still healthy, remain free of any infection and still suitable for the study.

If you do not receive the study virus when you attend for Quarantine, if you wish to (and are still eligible for the study) you may be able to come back for a later date (within 40 days from the last injection with the vaccine). You will be compensated for the amount of time you are in the Quarantine Unit.

We will take blood and urine samples and do a number of procedures and tests to check that you are suitable. These are described in **Section 8**.

We will ask you about your medical history and any medicines and treatments you have been taking.

If you remain well and are enrolled into the study, you will stay in your room in the Quarantine Unit for approximately 10 days. However, you may be discharged from the Quarantine unit later if you have been infected by the study virus and the virus can still be detected in your nose or if you are unwell.

You can bring things to keep you occupied, e.g., your mobile phone and laptop, and watch TV and films, but you cannot have any visitors.

In the Quarantine Unit staff will wear protective clothing and a hood covering their heads to prevent the spread of infection.

On Day 0, we will check you are still suitable to receive the study virus. If you are, you will be asked to lie flat on your back while the study nurse or study staff will place a few drops of the study virus




# INFORMED CONSENT FORM

solution into each of your nostrils. You will remain lying on your back for 10 minutes and the staff will continue to monitor you.

Over the course of the Quarantine period, we will do tests to check the effects of the study virus. Unfortunately, some procedures may have to be done during the night and early in the morning.

If you remain well and have 2 nasal swabs showing no study virus on 2 separate samples from different days you may leave the Quarantine Unit. However, you might be asked to stay longer if the study staff thinks it is necessary for safety reasons or if you still have an ongoing infection or positive nasal swab sample for study virus. When discharged, you will continue to record any symptoms you may still have into the Diary Card up until Day 35.

# 7.4 Visits 5 and 6: Follow-up

You will be required to return for 2 additional safety follow-up visits:

- > the first on day 35 (± 3 days), approximately 4 weeks after you leave guarantine, and
- > the second on Day 63 (± 5 days), approximately 8 weeks after you leave quarantine.

We will take blood and urine samples and do a number of procedures and tests that you will already have had during your stay in Quarantine, to check that you are well. These are described in **Section 8**.

We will ask you about your general medical health since discharge and any medicines and treatments you have been taking. The study staff will review and assess the completed self-testing records in the Diary Card during these visits.

If necessary, the study staff may ask you to come back again for another test, or be referred for further care should it be required.

# 8 Details of sampling and procedures we may perform

The following study procedures will be conducted according to the study schedule table on page 17:

- We will collect and test blood samples. During the Quarantine period, we may take several samples over a short time, so we may place a small plastic tube (cannula) into a vein in your hand or arm to make repeated sampling less painful. Placing a cannula in a vein, or taking blood using a needle can sometimes be uncomfortable, and could leave a bruise, or the vein could get inflamed or infected. These problems usually get better quickly, once the needle or cannula has been removed. Sitting or lying down when blood is taken should stop you feeling light headed or fainting.
- The amount of blood we collect will not exceed 470mL (about 1 pint the amount taken at a blood donation session) over a 5 month period. As a precaution, you should not give blood from 3 months prior to the anticipated date of first vaccination until 3 months after the last study visit.
- The study doctor will check your heart, breathing, ears, nose, throat, head and neck, lymph nodes (glands), abdomen, nerves, muscles, skin and eyes in a physical examination.
- Your height and weight will be measured.
- We will record your heart rate, breathing rate, blood pressure, and temperature, and we may check the amount of oxygen in your blood using a device temporarily clipped onto your finger.




# **INFORMED CONSENT FORM**

- We will collect and test urine samples to test for infection, ill health, drugs of abuse, and pregnancy (females only).
- We will carry out breath tests for alcohol.
- We will record an electrocardiogram (ECG) to look at your heart's activity. Small pads will be stuck to your arms, legs and chest (which may need to be shaved) while you lie still for a few minutes. The pads can sometimes cause minor skin irritation.
- We will also test your lung function using a 'spirometer'. You will take the deepest breath in you
  can, then exhale long and hard into a tube. This can make you cough or feel short of breath for
  a short time.
- We will take nasal swabs (i.e. cotton wool at the end of a small stick) using the procedure
  described below. Nasal sampling procedures can be uncomfortable for a few seconds, and can
  occasionally cause a nosebleed, make you sneeze, and/or leave you with watery eyes and a
  runny nose, but there are no long-term effects. We would advise you not to pick, rub or blow
  your nose too hard during the guarantine period.
  - A nasal 'swab' is put into each nostril to collect mucus and cells from the back of your throat behind your nose.
- After each injection with the study drug or placebo for around 3 weeks at home you will record your symptoms on a diary card which will be explained to you before you leave your appointment.
- During the Quarantine period and until Day 15 (at home), you will record your symptoms on a diary card.

# 9 Your responsibilities

Ask if you are unsure about anything.

Some of the important rules that you must follow are:

- You must tell the study staff if you take any medicines or treatments (e.g., tablets, sprays, creams, medicines and inhalers) that your GP/doctor told you to take, and/or any you have bought or obtained for yourself (e.g., multivitamins, homeopathic medicines). You will be told which medications are allowed during the study and which are not. During quarantine, you must not take any medications unless they have been given to you by the study doctor.
  - You must tell the study staff if you are currently a smoker, or have been in the past. The study staff will need to know the details about how much you smoke now, and have smoked in the past.
    - You will not be able to take part if you have ever smoked the equivalent of 10 pack years or more; one pack year is the equivalent of smoking 20 cigarettes (1 pack) every day for 1 year.
    - For those participants that are current casual smokers or use of smoking / nicotinerelated products, they must agree to refrain from smoking during the in-patient stay.
- Smoking and use of any nicotine-containing products (e.g., gum, nicotine patches, inhalers, e-


Version: Final v3.2 31JAN2017



# **INFORMED CONSENT FORM**

cigarettes) are not permitted in the hVIVO clinic or Quarantine. You must agree not to smoke while at hVIVO premises.

- You must tell the study staff approximately how much alcohol you currently drink. You must not consume any alcohol for at least 1 day before you receive your first dose of study vaccine, admission to quarantine, throughout quarantine, and 1 day before each follow-up visit. This includes alcohol contained in both drinks and food.
- Please note that only decaffeinated drinks are provided in the Quarantine Unit.
- You must not use 'legal highs' and drugs such as amphetamines, benzodiazepines, cocaine, cannabinoids, barbiturates, opiates, and methadone from screening until after the last study follow-up visit. Any recent history of abuse of the above drugs with a positive urine test could result in your exclusion from the study. Please avoid the use of codeine and any food items containing poppy seeds for at least 7 days before your screening visit and for the duration of the study.
- You must not become pregnant or get someone pregnant during the study and for 90 days afterwards. (see Section 10.3 'Potential harm to an unborn child'). The study staff will advise you appropriately.
- Women who are breastfeeding or pregnant cannot take part in this study.
- You should avoid energetic physical activity for at least 3 days before you are admitted to quarantine until after the last study follow-up visit. Unaccustomed or energetic exercise may result in abnormal blood test which could result in your being excluded from the remaining part of the study.
- If you have any insurance policies, you should check whether taking part in this research study affects them.

If you do not cooperate with the study procedures, we may withdraw you from the study, which could lessen the amount of compensation you get (see Section 13).

# 10 What are the possible drawbacks of taking part?

The known effects of the study virus and study vaccine are described below, however, there may also be unexpected risks related to the study virus, the study vaccine and study procedures. While you are in the Quarantine Unit the medical staff will monitor your condition closely, and medical assistance will be available at all times. You must tell us immediately if you have any symptoms or changes in your wellbeing.

We will tell you as soon as possible if we become aware of new information that could change your mind about taking part in the study.

If we find any abnormalities at screening or during the study, we will inform your GP or a specialist if necessary, after discussing them with you.

# 10.1 Effects of the study virus

After inoculation with the study virus, you might experience symptoms of influenza. In healthy adults, the illness usually resolves within a week with relief of symptoms occurring naturally within two weeks.

From two days before the planned discharge day, consecutive day nasal swabs will be tested for the




# INFORMED CONSENT FORM

study virus, and you will only be allowed to leave if you are considered to be well enough and not likely to infect other people.

As a precaution, for 2 weeks after you leave the Quarantine Unit, you should avoid close contact with anyone who could become very ill if they were to be infected with the study virus, e.g., children under 5 years old, anyone who lives in a nursing home, anyone with a low resistance to infection or who takes drugs that lower their resistance, anyone who is having or is about to have drug treatment for cancer (chemotherapy), and anyone who has chronic obstructive pulmonary disease (COPD), emphysema or other severe lung disease, or who has had a bone marrow or solid organ transplant.

If you are a healthcare worker, nurse, doctor, or medical student, you should not work with patients until 2 weeks after you leave the Quarantine Unit, or until any symptoms are fully resolved (whichever is the longer period).

Although the risk of passing on the virus is very small, Influenza infections can cause complications in pregnant women, therefore male subjects who have a partner that is pregnant or likely to become pregnant during the study should not take part

# 10.2 Side effects of study drug

So far the study vaccine has demonstrated an excellent tolerability and safety profile in both animal studies and in 2 early clinical studies in healthy volunteers.

When this study starts the study vaccine would have been given to 56 subjects in clinical trials at a similar dose level, with or without adjuvant (ISA-51). Results to date indicate that the study drug is generally well tolerated in humans, without significant adverse effects. The adverse events seen most frequently have been mild to moderate reactions and include:

Local reactions: bruising, pain at injection site, redness, swelling, itches.

Systemic reactions: chills, fever, malaise, muscle pain, joint pain, nausea, headache, sweating, tiredness.

For the adjuvant given with the vaccine the most common expected local reactions are pain, redness, tenderness or swelling. Systemic reactions include: joint & muscle pain, chills, fever, headache, nausea, and tiredness.

The intensity is usually mild to moderate and usually transient.

Should this information change once the full study results are available you will be provided with the new information and asked to provide additional consent to confirm your willingness to take part. If you do not understand what any of these side effects mean, please ask the study staff to explain these terms to you.

You may have an allergic reaction to the study vaccine. Symptoms of an allergic reaction may include the following; headache, rash, flushing, swelling, shortness of breath, nausea, and vomiting.

You will be closely monitored for any side effects.

There may also be other side effects that we are not yet aware of, so you must tell us immediately if you have any symptoms or changes in your wellbeing.

# 10.3 Potential harm to an unborn child

The following contraceptive requirements apply to all participants who receive the experimental




# **INFORMED CONSENT FORM**

vaccine, stay in Quarantine and receive a virus.

The effect of the study vaccine on reproduction and an unborn child are unknown, and it is possible that the study vaccine could harm an unborn baby. Therefore, only women who are not pregnant and are of non-childbearing potential may participate. We will do pregnancy tests at screening and during the study.

In this study, to be of 'non-childbearing potential' a woman must either have documented proof of surgical sterilisation or hysterectomy, or be post-menopausal. Post-menopausal is defined as having had 24 months of complete absence of menstrual periods (amenorrhea), and post-menopausal levels of Follicle Stimulating Hormone (FSH). Post-menopausal women cannot be using hormone replacement therapy (HRT).

Female partners of male subjects must not be pregnant or become pregnant during the study and for up to 90 days after the male subject has completed the study.

Both men (and their female sexual partners) and women who participate in this study must use acceptable methods of birth control throughout the course of the entire study and for 90 days after completion of the study. If you are a man whose female sexual partner becomes pregnant within 90 days after completing this study, the study staff will need to follow up regarding your partner's pregnancy and your child's health.

Male subjects must use a male condom with spermicide.

In addition, a female subject or partner must use one of the following methods of contraception: established (i.e., a minimum of 2 weeks prior to admission) use of a non-hormonal intra-uterine device (IUD) with spermicide, female condom with spermicide, contraceptive sponge with spermicide, diaphragm with spermicide, cervical cap with spermicide, or oral, implantable, transdermal, or injectable contraceptives (plus a barrier method). Periodic abstinence (e.g., calendar, ovulation, symptothermal and post-ovulation methods) and withdrawal are not acceptable methods of contraception.

Male and female condoms should not be used at the same time due to risk of tearing.

Males must not donate sperm for 90 days after completing the study. Please share this information with your partner and talk to the study staff to decide the best method of birth control.

# 11 What if something goes wrong?

You must tell the study staff immediately if you have any health problems during the study. You will be given an emergency contact card after receiving the first vaccine, which provides a 24 hour telephone service in case you need to contact us outside of office hours. If you are injured or become unexpectedly sick as a result of taking part, hVIVO will offer you the appropriate treatment. If you suffer any significant deterioration in health or well-being caused directly by participation in the study, compensation will be paid by the Sponsor in accordance with the Association of the British Pharmaceutical Industry (ABPI) guidelines. Further information regarding the mentioned guidelines is available request **hVIVO** the internet (http://www.abpi.org.uk/ouron or on work/library/guidelines/Documents/compensation guidelines 2014.pdf) Please do not hesitate to ask for a copy of this guideline from hVIVO, if you wish to read it.

By agreeing to take part in this study, you do not give up any legal rights to other treatments that may be available to you for an injury or illness caused by the study drug or study procedures.




# INFORMED CONSENT FORM

# 12 Could my participation end early?

hVIVO or Sponsor can stop the study at any time and the study doctor could withdraw you if he/she thinks it is in your best interests.

If you decide to withdraw and have already been given the study virus, you will be advised to stay in the Quarantine Unit until you cannot infect other people, and also to attend for a follow-up visit so that your condition can be assessed. We may ask you to have some health tests.

If you withdraw from the study you will be asked to sign a form telling us how you would like us to deal with your study samples and information. You can choose either 'No further participation' or 'No further use of my samples or data'.

You may be advised to attend for a follow-up visit so that your condition can be assessed. We may ask you to have some health tests to confirm you are well.

'No further participation' means that hVIVO would still have your permission to keep and use any data and samples you have already provided, but no more samples or data would be collected or analysed.

'No further use of my samples or data' means that hVIVO would destroy your samples; and your data and samples would not be used in any future analyses.

In both cases, you may also ask hVIVO to remove your personal details (e.g., address and date of birth) from its participant database. However please note, it would not be possible to withdraw your data from analyses that have already been done as hVIVO need to keep and use any research data already collected, in order to comply with their legal obligations and to maintain the scientific integrity of the study.

A record of your signed consent and your withdrawal would be kept as a record of your wishes.

# 13 Expenses and compensation for taking part

You will be compensated for your participation in the study as follows:

Attendance at the Screening visit:

 £100 (for time and travel expense) will be paid shortly (i.e., within about 2 weeks) after the Screening visit.

If you complete the full Quarantine phase and the follow-up visit at Day 63 ( $\pm$  5 days), you will receive a total of £3000. This total (which includes reasonable travel expenses to and from the Quarantine Unit) will be split into 4 payments:

- £250 will be paid shortly after first vaccination
- £250 will be paid shortly after second vaccination
- £1000 will be paid shortly after the end of Quarantine.
- £1500 will be paid shortly after the Day 63 (± 5 days) follow-up visit.

Additional visits or expenses:

If you are asked to attend for additional visits, reasonable time and travel expenses will be reimbursed for each visit at the hVIVO's discretion. Compensation in the event of withdrawal or exclusion:




# **INFORMED CONSENT FORM**

- If you withdraw or are excluded from Quarantine before the virus is administered, you will receive
  a total of £200 approximately 30 working days after leaving Quarantine.
- If you withdraw or are excluded from Quarantine after the virus is administered, you will be compensated for each day in the Quarantine facility at pro rata rate, in addition to the screening payment, approximately 30 working days after leaving Quarantine.

hVIVO will not pay tax or National Insurance from the money due to you. It is your responsibility to pay these. Contact HM Revenue & Customs for information (<a href="http://www.hmrc.gov.uk/">http://www.hmrc.gov.uk/</a>) or telephone 0300 200 3300).

Please note that there are some situations where we are required to tell the authorities about your payments if we are asked to.

# 14 Future contact with hVIVO

hVIVO may contact you after your participation in this trial. If analysis of your data proves to be of particular interest to researchers, you may be contacted and invited back to hVIVO to provide further consent and samples/data. For example, you may be of interest to researchers if you are given a virus but do not become infected.

# 15 Participation in other research studies

You should not take part in too many clinical trials, or in several clinical trials at the same time. Research units like hVIVO keep a linked database of research participants in which your National Insurance number, or passport number and country of origin are recorded along with the dates you were given a virus, and if you have taken part in a drug trial. Your details are kept for at least 2 years. We will check the database before you join a clinical trial, and if necessary, we may be able to trace you through it.

# 16 Storage and use of samples and information from this research

hVIVO will send your samples for testing in our laboratories where they will be stored securely within the hVIVO Research Tissue Bank until they are unusable or finished. Your samples and information will be labelled, but we will not use your name or information that could identify you.

hVIVO may send some of your samples to research laboratories in other European countries and the United States of America (USA), and to other parties for research. Any movement and storage of samples will be in accordance with the Human Tissue Act 2004 and other relevant laws in the countries they are sent to. hVIVO will own all the samples and related data collected from you during your participation in a clinical trial, and the rights comprised in or related to such samples or data.

At the end of this research study, it is very likely that we will have some samples left over that were not required for the tests. This is because all research studies collect sufficient sample volumes to allow for repeat testing in case the laboratory tests fail. Spare samples that were not needed could be useful to other researchers for future research.

hVIVO has been given permission under the UK Human Tissue Act 2004 (UK law) to store such samples securely at its licensed hVIVO tissue bank (located at hVIVO premises) until the ethically approved testing of the stored samples has been performed. We will ask you to give your consent for this if you want to participate in this study. If you give your consent to this, your leftover samples and their related information from this research study will be stored and used for further research that has




# **INFORMED CONSENT FORM**

been ethically approved. You would not be told the results of such research.

# 17 Will my taking part be kept confidential?

hVIVO will keep your information (including your results and data) in paper records and in computer databases. hVIVO staff involved in the collection, processing or storage of your personal data are trained on how to handle data. You will not be identified personally in any publication or presentation about the research. hVIVO will keep your information for at least 5 years.

hVIVO may share your personal and medical information with partners, or those working with partners that have facilities in other countries, including countries outside the European Economic Area (EEA) and the USA. Some use of this information may take place in countries with lower data protection standards than the UK. By signing the Informed Consent Form, you agree to any such transfer, use or storage of information outside of the UK, and outside the EEA. hVIVO's partners will ensure that information transferred outside your country of residence is treated in accordance with the content of the Informed Consent Form.

hVIVO and/or its representatives, independent auditors, government representatives and the Research Ethics Committee (REC) may need to check your medical and research records. Your information and samples may also be used in other research into respiratory viruses but this will always be in line with the law.

In the hVIVO premises, for safety reasons, shared areas are monitored using closed-circuit television (CCTV), which is only seen by hVIVO staff and their clients, and occasionally by people inspecting our facilities and/or research processes. The CCTV is located in public places only, not pointing into your room. The CCTV does not give sound and is not stored electronically or on tapes. You will not be named in any images although somebody could recognise your face. Additionally, we may want to take digital photographs or videos of you alone or in a group, to use for staff training, and to show what we do at hVIVO. Although the copyright in these images will belong to hVIVO, the images will only be used in line with UK data protection laws. You will not be named in any pictures, although someone could recognise your face. You may ask for a copy of any photos or video recordings you appear in. If you do not wish to appear in a photograph or video then you can choose not to and let us know. You can still take part in the study even if you do not want to be in any photographs or videos. If you agree, then change your mind, the photographs will be destroyed or deleted, and your image will be blurred out in any videos.

Please ask the hVIVO staff if you have any questions about the way your information is collected and used. Data protection laws give you certain rights that allow you to have access to data held about you (and if needed, correction of such data), and the right to object or prevent certain processing of your information if it could cause you harm or distress. You may obtain access to such data by contacting hVIVO (see Section 20 'Contact for questions or complaints').

If you want to know more about your rights and how you can enforce them, please contact the Information Commissioner (at Wycliffe House, Water Lane, Wilmslow, Cheshire, SK9 5AF. (<a href="http://www.ico.gov.uk">http://www.ico.gov.uk</a>), or telephone 0303 123 1113 (local rate) or 01625 545745 (national rate).

#### 18 Who has approved this research?

North East – York Research Ethics Committee has looked at the details of this study and has given its approval for the study to go ahead. If you have any questions about your rights as a participant in




# **INFORMED CONSENT FORM**

this study, you can contact the REC on 0207 104 8084.

# 19 Research registry

A description of this study and a summary of the results will be available on several clinical trial databases [e.g. http://www.ClinicalTrials.gov]. This will not include information that could identify you.

# 20 Contact for questions or complaints

If you have any questions about taking part in this research, contact a member of hVIVO staff on 020 7756 1414, or Freephone 0800 756 6334. If you believe that you suffered an injury as a result of taking part in this research, contact a member of hVIVO staff on 020 7756 1414, or Freephone number 0203 126 4029.


Version: Final v3.2 31JAN2017



# **INFORMED CONSENT FORM**

Protocol Title: Phase IIb Study of the Efficacy of Flu-v, a Broad Spectrum Influenza

Vaccine in an H1N1 Influenza Healthy Human Challenge Model

Protocol number: FLU-v-004

Protocol version: Final v2.2\_31JAN2017

Research Ethics

Committee (REC)

16/NE/0227

Ref:

EudraCT Number: 2016-002134-74

Sponsor: PepTcell Limited (t/a SEEK)

**SEEK** 

Central Point,

Sponsor's address: 45 Beech Street,

London, EC27 8AD

Principal Investigator: Dr Andrea Guerra

Research sites: hVIVO Services Limited (hVIVO) sites at:

Queen Mary BioEnterprises Innovation Centre

(1) 42 New Road, London E1 2AX, UK

Telephone: 0207 756 1414 Manchester Science Parks

(2) Kilburn House, Lloyd Street North Manchester M15 6SE, UK

Telephone: 0161 402 3470

Dr Jeremy Dennison

Pharmacy and clinical services

(3) Hammersmith Medicines Research Ltd

Cumberland Avenue, London, NW10 7EW, UK

Telephone: 0208 961 4130

| Participant No: | | Participant's<br>Name: → | | | | |
|---|---|---|---|---|---|---|
| | | | First name | Middle name | Last na | ame |
| Please read the following statements about your consent to take part in this research and | | | | | | |
| initial the boxes alongside to confirm your consent. To take part, you must confirm your | | | | | | |
| consent for all points (1-10 inclusive). | | | | | | |
| 1. | I have read and understood Final Version 3.2 of the Participant Information Sheet dated 31JAN2017 for the above-mentioned research. I have had the opportunity to ask questions, I have had these answered to my satisfaction, and I have had enough time to consider my participation. | | | | | |
| 2. | I understand that taking part is voluntary, and that I am free to withdraw at any time without giving a reason, and without my medical care or legal rights being affected. | | | | | |
| 3. | I agree to my GP or doctor being informed of my participation and to the provision of a copy of my medical records to hVIVO. I agree to allow hVIVO to share my results with my GP or doctor if required. | | | | | |


**Protocol Number**: FLU-v-004 **Version**: Final v3.2\_31JAN2017



# **INFORMED CONSENT FORM**

| | IN ORMED CONSENT FORM | |
|---|---|---|
| 4. | I understand that my blood will be tested for Human Immunodeficiency Virus (HIV), and Hepatitis A, B and C viruses. I have been told about the consequences of a positive result, and the effect this could have on employment and any life assurance and health insurance policies I may have. I understand that I must have negative HIV, Hepatitis A, B and C results to take part in the study. I give consent for my blood to be tested for HIV, and Hepatitis A, B and C viruses; and for my GP to be informed if I test positive for any of the viruses outlined above. | |
| 5. | I understand that relevant sections of my medical notes and data collected may be looked at by individuals from hVIVO, independent auditors, its representatives, regulatory authorities, where it is relevant to my taking part in this research. By signing this consent form, I give permission for these individuals to access my medical records. | |
| 6. | I understand the possible risks of passing the virus to vulnerable people after discharge from the Quarantine Unit, as described in the Participant Information Sheet. | |
| 7. | I understand that data protection laws differ in non-EEA countries and if I do not want my anonymised data to be sent outside of the EEA, I will not be able to take part in this study. I agree that my samples and anonymised data <u>can</u> be sent outside of the EEA. | |
| 8. | I assign all rights in the samples, related data and materials I provide to hVIVO, and acknowledge that hVIVO will own such materials and the rights in them, even after my incapacity or death. | |
| 9. | I agree to the samples and procedures detailed in the Participant Information sheet above. | |
| 10. | I agree to take part in the above mentioned research. | |
| Please i | nitial each of the following boxes to indicate that you have read and understood each | n of the |
| following | g statements, then circle either YES or NO to indicate your choice. | |
| 11. | I understand that I have the choice to allow hVIVO to store and use my leftover samples and data for future health research and laboratory method and equipment testing. My samples will be handled according to ethical standards, and where required, subject to ethical approval. I understand that I will not be informed of any details of my health status that may be discovered by future research using my samples or information. I agree to allow my leftover samples and data to be used by hVIVO for future health research and for laboratory testing. YES NO (Please circle) | |
| 12. | I understand that I have the choice to allow hVIVO's research partners to store and use my leftover samples and data for future health research and laboratory method and equipment testing. My samples will be handled according to ethical standards and where required, subject to ethical approval. I understand that I will not be informed of any details of my health status that may be discovered by future research using my samples or information I agree to allow my leftover samples and data to be used by hVIVO's research partners for future health research and for laboratory testing. YES NO (Please circle) | |
| 13. | I understand that digital photographs and video recordings may be taken in Quarantine. If I agree, I may have a copy of pictures containing my image, and I may ask for my image(s) to be removed or destroyed if I withdraw my consent to this photography and video recording. I understand that I can still participate if I do not agree to this. I give my consent to be included in digital photographs and videos recordings. YES NO (Please circle) | |




# **INFORMED CONSENT FORM**

| 14. | I have been informed that noiseless CCTV is used in public areas in the hVIVO clinic and Quarantine Unit, but images are not recorded. |
|---|---|
| | YES NO (Please circle) |
| 15. | I give my consent for hVIVO to contact me in the future. |
| | YES NO (Please circle) |
| 16. | I understand that I have the choice to allow hVIVO to store any viruses that are |
| | found in my samples during this study for further research use. |
| | YES NO (Please circle) |

| Please indicate your consent by completing the box below | | | | |
|---|---|---|---|---|
| ▼ THIS PART TO BE COMPLETED BY THE PARTICIPANT | | | | |
| | | | ) MMM YYYY | HH: MM |
| Participant's signature | Da | te | Time | |
| ◆ PARTICIPANT'S FULL NAME IN BLOCK CAPITALS ◆ | | | | |
| PARTICIPANT'S FIRST NAME | MIDDLE NAME | LAST NAME | | |
| ♥ THIS PART TO BE COMPLETED BY THE PHYSICIAN (OR DELEGATE) OBTAINING CONSENT ♥ | | | | |
| | DD MMM YYYY | | YY HH: | MM |
| Physician's (or delegate's) signature | Date | | Time | ) |
| ♥ PHYSICIAN'S (OR DELEGATE'S) NAME IN BLOCK CAPITALS ♥ | | | | |
| PHYSICIAN'S (OR DELEGATE'S) FIRST NAME | MIDDLE NAME | LAST NAME | | = |

